CLINICAL TRIAL: NCT04428463
Title: Fibrinogen- Based Collagen Fleece Graft Myringoplasty for Chronic Tympanic Membrane Perforations - a Prospective Study
Brief Title: Repair of Tympanic Membrane Perforation Using Tachosil Under Local Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMC-13-20
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Tympanic Membrane Perforation
Keywords: tympanic membrane perforation; tachosil; local anesthesia
MeSH Terms: conditions — Tympanic Membrane Perforation | interventions — TachoSil

STUDY DESIGN:
Intervention Model Description: two groups. In one we will use the conventional treatment strategy using tympanoplasty with fascia and cartilage.
  in the intervention group we will use tachosil in closing the perforations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tympanoplasty using fascia and cartilage (Active Comparator): tympanoplasty under general anesthesia using fascia and cartilage witch is the gold standard for treating tympanic membrane perforations.
  Interventions: Procedure: fascia and cartilage
- Tachosil (Experimental): repair of tympanic perforations under local anesthesia using Tachosil patch.
  Interventions: Procedure: Tachosil

INTERVENTIONS:
Procedure: Tachosil — tympanic membrane perforation repair using Tachosil patch under local anesthesia
  Arms: Tachosil
Procedure: fascia and cartilage — tympanic membrane perforation repair using fascia and cartilage under general anesthesia
  Arms: tympanoplasty using fascia and cartilage

SUMMARY:
Tympanic membrane perforations are common medical problem that encounters a lot of patients in all age groups.

The gold standard for treatment of perforations is tympanic membrane closure procedure (tympanoplasty) which is done under general anesthesia.

This procedure could be problematic for many patients who are not suitable for general anesthesia due to their medical status.

It's also time consuming for the patient and for the medical system, since it takes a lot of time to reach the operation room and hospitalization for at least two days.

The purpose in this study is to use Tachosil (Fibrinogen based patch) under local anesthesia to close tympanic membrane perforations.

Tachosil is in use for hemostasis and for tissue repair after injury. Tachosil is bound to the tissue and form a waterproof membrane. In the setting of ENT clinic and under local anesthesia, the investigators will start the procedure with debridement of the tympanic perforation edges, then they will close the perforation using two pieces of Tachosil under and above the perforation in the right form (active side to the active side).

If the results will be similar to tympanoplasty results, this method may be used for closure of tympanic perforation and save time and money for the patient and for the health system.

DETAILED DESCRIPTION:
Tympanoplasty is the gold standard treatment for tympanic membrane perforation.

It is done under general anesthesia in the following form:

Incision in the post auricular area, harvesting of fascia and cartilage from the concha of the pinna .

In Trans ear canal approach starting with debridement of the edges of the tympanic membrane perforation and closing the perforation using cartilage and fascia.

After being informed about the study and potential risks, all patients giving informed consent will participate in the study.

This study will include two groups. The first group will be treated with the conventional way as described above. The interventional group will be treated using Tachosil in the following order:

Local anesthesia using Lidocadren (lidocaine and epinephrine) will be injected to the ear canal using dental needle.

Debridement of the edges of the tympanic membrane perforation Placing the tachosil under and above the perforation in the correct order. The patient could be discharged home immediately after the procedure if no adverse effects are seen (dizziness, nausea or vomiting).

After one month, similar to the conventional treatment method, the patient will be invited to the otology clinic, for hearing test and microscopic examuntaion of the tympanic membrane, to see if the perforation is closed.

The study will compare the success rate in the two groups and if it will be similar that will help publish this method and use it in patients who are not suitable to general anesthesia and in hospitals were waiting time table for operation room is very long.

ELIGIBILITY:
Inclusion Criteria:

* chronic tympanic membrane perforation
* dry ear at least 4 weeks before the procedure
* no evidence of cholesteatoma
* hearing test in the last 3 months
* signing informed consent

Exclusion Criteria:

* age under 18 years
* pregnant
* breastfeeding
* a known sensitivity for any ingredient
* a perforation that is more than one third of the tympanic membrane area.
* new onset perforation (less than 3 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2020-06-30 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
closure of tympanic membrane perforation | one month after the procedure
  one month post operative the patient will be re-examined in the clinic to see if the perforation is closed.